CLINICAL TRIAL: NCT00813007
Title: Radical Trachelectomy for Women With Early Stage Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0723
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Cervix; Questionnaire; Adenocarcinoma of uterine cervix; Squamous cell carcinoma of uterine cervix; Adenosquamous carcinoma of uterine cervix; Abdominal radical trachelectomy; Trachelectomy; Quality of life; Sexual functioning
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire: Radical trachelectomy outcomes for cervical cancer
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — 5 Questionnaires at differing times before and after surgery.
  Other Names: Survey

SUMMARY:
The goal of this research study is to learn about quality of life, sexual functioning, and symptoms in women who have undergone abdominal radical trachelectomy for cervical cancer.

This is an investigational study.

Up to 100 patients will be enrolled in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Before Surgery:

If you agree to take part in this study, before you have the abdominal radical trachelectomy surgery, the following information will be recorded during one of your regular clinic visits:

* Your race and date of birth.
* Your complete medical and surgical history, including the date of your diagnosis and your diagnosis before surgery.
* Your weight, height, and body mass index.

During and After Surgery:

During and after surgery, the following information will be gathered from your medical record or you will be asked:

* If there was any blood loss during surgery.
* How long the surgery lasted.
* If there were any complications during the surgery.
* If you needed any blood transfusions.
* What type of instrument was used for preventing or sealing blood loss.
* How long you stayed in the hospital.
* If you experienced any infections within 1 month after surgery.
* If you experienced any complications within 1 month or later than 1 month after surgery.
* The length of time it took to recover your bowel and urinary function.
* If you received any treatments for cancer after surgery, such as radiation therapy, chemotherapy, or hormonal therapy.

Once a year for up to 5 years, if you return for an annual routine follow up visit, the results of any pap smears you have had will be collected.

Once a year for up to 5 years, you will also be asked the following questions about your health and fertility, either by mail or during a regular clinic visit:

* What is the status of the disease?
* Did you want to get pregnant in the last year?
* Did you attempt to get pregnant?
* Did you become pregnant? If so, how you became pregnant and the outcome of the pregnancy? If not how long did you try to become pregnant and did you try any form of assisted reproduction?

Questionnaires:

You will complete 4-5 questionnaires at each of the following times:

* Within 2 weeks before your surgery.
* At 4-6 weeks after surgery
* At 6 months after surgery.
* At 1 year after surgery.
* Once a year for the next 4 years.

These questionnaires will ask about your physical health, mental and emotional health, pain, vitality, social functioning, general health, quality of life, and sexual functioning. It will take about 15 minutes to complete 5 questionnaires. If you do not receive your follow-up care at MD Anderson, the questionnaires will be mailed to you at the above time-points with a prepaid return envelope. Mailed questionnaires will be returned to the study chair in an envelope marked CONFIDENTIAL with NO RETURN ADDRESS on the return envelope. Your name will not appear on the questionnaires or return envelope. Instead, a code will be used (on the questionnaires only) that will connect the questionnaires with your medical record. Only the study chair or study coordinator will have access to the code document. The document is kept in a locked filing cabinet and/or password protected computer. All responses will be stored in a locked office.

Length of Study:

You will be on study for up to 5 years. If the disease returns, you will be taken off study.

ELIGIBILITY:
Inclusion Criteria:

1. Women with histologically confirmed, primary adenocarcinoma, squamous cell carcinoma or adenosquamous carcinoma of the uterine cervix
2. Patients with FIGO stage IA1 (with lymph vascular space invasion), IA2, or IB1 disease
3. Patients must be suitable candidates for surgery
4. Patients who have signed an approved Informed Consent
5. Patients with a prior malignancy allowed if > 3 years previous with no current evidence of disease
6. Females older than 18 years who are undergoing radical trachelectomy
7. Women must be able to read and write in either Spanish or English

Exclusion Criteria:

1. Any histological type other than adenocarcinoma, squamous cell carcinoma or adenosquamous carcinoma of the uterine cervix
2. Tumor size greater than 4 cm
3. FIGO stage II-IV disease
4. Patients with a history of pelvic or abdominal radiotherapy
5. Patients who are pregnant
6. Patients with contraindications to surgery
7. Patients with evidence of metastatic disease by conventional imaging studies, enlarged pelvic or aortic lymph nodes > 2cm; or histologically positive lymph nodes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with histologically confirmed, primary adenocarcinoma, squamous cell carcinoma or adenosquamous carcinoma of the uterine cervix.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-12-16 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean scores for the General Health-Related Quality of Life (SF-12) | Follow up visits annually
  Completed SF-12 questionnaires at baseline and at each follow-up visit (4-6 weeks, 6 months, 1 year, and annually for 4 more years)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Frumovitz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org